CLINICAL TRIAL: NCT06201325
Title: Comparison of the Effectiveness of Virtual Reality Based Exercises and Conventional Physical Therapy in the Treatment of Adhesive Capsulitis
Brief Title: The Effects of Virtual Reality Based Exercises in Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, medical doctor, assistant prof, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-19/146
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis; virtual reality; conventional physical therapy
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Patients will be randomly divided into 3 groups. They will be selected by simple random sampling using the closed envelope method.
  In the first group, will be included in a VR-based exercise program for half an hour a day, 5 days a week for a total of 3 weeks, in addition to home exercise programs for half an hour a day, 5 days a week for a total of 3 weeks. These individuals will use the Microsoft Kinect for Azure VR system in the virtual environment.
  In the second group, will be included in the traditional exercise group, will be included in the stretching and strengthening exercise program for half an hour a day, 5 days a week for a total of 3 weeks, in addition to home exercise programs for half an hour a day, 5 days a week for a total of 3 weeks.
  In the third group, who will be included in the home exercise group, exercises will be taught to the patient and will be applied for half an hour a day, 5 days a week for a total of 3 weeks.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assesor will be different persons
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR group (Active Comparator): VR-based exercise program for half an hour a day, 5 days a week for a total of 3 weeks, in addition to home exercise programs for half an hour a day, 5 days a week for a total of 3 weeks. These individuals will use the Microsoft Kinect for Azure VR system in the virtual environment. They will play the registered games. These games will include purpose-oriented activities such as lying on the shelf and using bilaterally, which are intended to use the upper extremities of individuals with AC in daily life.
  Interventions: Other: virtual reality based exercises; Other: home exercises program
- Conventional group (Active Comparator): Individuals in the second group, who will be included in the traditional exercise group, will be included in the stretching and strengthening exercise program for half an hour a day, 5 days a week for a total of 3 weeks, in addition to home exercise programs for half an hour a day, 5 days a week for a total of 3 weeks. The exercises will be performed by a physiotherapist working in the clinic and blind to the study.
  Interventions: Other: conventional physical therapy; Other: home exercises program
- Control group (Other): In the third group, who will be included in the home exercise group, exercises will be taught to the patient and will be applied for half an hour a day, 5 days a week for a total of 3 weeks.
  Interventions: Other: home exercises program

INTERVENTIONS:
Other: virtual reality based exercises — play VR games
  Arms: VR group
Other: conventional physical therapy — streching and strengthening exercises
  Arms: Conventional group
Other: home exercises program — home exercises

SUMMARY:
The aim of this study is to evaluate the effectiveness of virtual reality based exercises and conventional physical therapy on shoulder pain, mobility, functional ability and quality of life in adhesive capsulitis and to investigate whether it is superior to the control group.

DETAILED DESCRIPTION:
Adhesive capsulitis(AC) is an enigmatic condition characterized by painful, progressive and disabling loss of active and passive shoulder joint range of motion in multiple planes. Approximately 2% to 5% of adults between age 40 and 70 develop adhesive capsulitis with a greater occurrence in women and in individuals with thyroid disease or diabetes. AC is an arthroﬁbrosis involving the formation of excessive adhesions along the glenohumeral joint. It is a disease of unknown aetiology and is classified as primary and secondary. Primary adhesive capsulitis includes cases of idiopathic origin resulting from chronic inﬂammation with ﬁbroblast proliferation. Secondary adhesive capsulitis includes central nervous system problem, prolonged immobilisation of the arm, trauma or fracture, infectious diseases, etc. The progression of adhesive capsulitis is characterised by four stages, each stage showing a distinctive clinical presentation:

1. Painful phase: lasts less than three months and is characterised by shoulder pain at night with preserved glenohumeral motion.
2. Freezing phase: lasts three to nine months and is characterised by severe pain and stiffness in the glenohumeral joint.
3. Frozen shoulder process: lasts nine to fourteen months and is characterised by loss of movement and pain in all directions at the end.
4. Thawing phase: lasts fifteen to twenty-four months and is characterised by persistent stiffness, minimal pain, delayed recovery of shoulder movement.

Interventions for this pathology usually include physical therapy, nonsteroidal anti-inflammatory drug therapy, intra-articular steroid injections, distension arthrography and surgery. Physical therapy is the mainstay of treatment for patients with adhesive capsulitis. Conventional physical therapy consists of electrotherapy modalities such as TENS, Interferential current, Ultrasound, low intensity laser and exercises such as stretching exercises, Codman Exercise, Wand exercises and joint mobilisation and is used to control pain, increase flexibility and improve range of motion.

It is known that it takes a long time to achieve pain relief and a good improvement in ROM in adhesive capsulitis. This situation affects the quality of life of patients and creates a need for easily accessible treatment options that provide faster recovery.

One of the main challenges facing the therapist in the treatment of adhesive capsulitis is to motivate the patient throughout conventional therapy. As noted in a recent review, individuals are more interested in leisure activities rather than performing repetitive tasks during therapy. Virtual reality (VR) is a three-dimensional computer-aided programme built with a system that creates virtual reality movements and generates a high amount of visual and sensory feedback during exercise. As a result, virtual reality (VR) has been used in many medical indications and has been shown to promote adherence to treatment by increasing patient motivation.

Different VR systems have been shown to be effective in individuals with kinesiophobia as well as stroke patients. Virtual reality guided exercise is a proven method already used in stroke, Parkinson's, cerebral palsy rehabilitation, vestibular rehabilitation and orthopaedic rehabilitation. However, there is limited data on its effectiveness in patients with adhesive capsulitis. This randomized controlled study will contribute to the literature by investigating the effects of VR based exercises in individuals with AC.

The estimated number of volunteers expected to participate in the study was determined according to power analysis. The sample size of the study was determined by the GPower 3.1.9.7 program, and by using the finding in a similar study in the literature, it was used with 80% power and 5% margin of error to catch the medium effect size between dependent measurements. It was decided to work with a total of minimum 60 people, 20 in each group. Considering the patients who may be excluded from follow-up in the study, it is planned to start the study with 75 patients. The diagnosis of the disease will be made by history and clinical physical examination and no additional imaging technique will be required.

Patients will be randomly divided into 3 groups. They will be selected by simple random sampling using the closed envelope method, and then Group A (virtual reality + home exercise ), Group B (conventional therapy+ home exercise ) and Group C ( only home exercise ).

Individuals in the first group to be included in the study group will be included in a VR-based exercise program for half an hour a day, 5 days a week for a total of 3 weeks, in addition to home exercise programs for half an hour a day, 5 days a week for a total of 3 weeks. These individuals will use the Microsoft Kinect for Azure VR system in the virtual environment. They will play the registered games. These games will include purpose-oriented activities such as lying on the shelf and using bilaterally, which are intended to use the upper extremities of individuals with AC in daily life. Participants will be treated under the constant supervision of a physiotherapist, will be rested at the end of the exercise, and will leave the clinic after making sure that there is no problem.

Individuals in the second group, who will be included in the traditional exercise group, will be included in the stretching and strengthening exercise program for half an hour a day, 5 days a week for a total of 3 weeks, in addition to home exercise programs for half an hour a day, 5 days a week for a total of 3 weeks. The exercises will be performed by a physiotherapist working in the clinic and blind to the study.

Individuals in the third group, who will be included in the home exercise group, exercises will be taught to the patient and will be applied for half an hour a day, 5 days a week for a total of 3 weeks.

The home exercise programme will be demonstrated by the physiotherapist at the beginning of the treatment and all groups will be asked to perform these exercises at home. Patients will be given a chart and they will be asked to mark this chart on the day they exercise. The exercise compliance of the patients will be monitored with this chart.

Home exercises will be organised as pendulum (Codman), finger ladder, Wand exercises, towel stretch and will be given to the patient as a visually printed exercise sheet.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65
* Clinical diagnosis of adhesive capsulitis
* Patients with loss of range of motion in a capsular pattern (external rotation >abduction > internal rotation)
* Participant signed informed consent

Exclusion Criteria:

* Surgery on the upper extremity or trunk
* Upper extremity injury in the last 6 months
* Injections in the shoulder area in the last 6 months
* Systemic or local infection of shoulder
* Uncontrolled hypertension
* Inability to cooperate VR
* Patient with malignancy
* Neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 0( baseline)
  The Visual Analog Scale is a pain rating scale with the numbers 0. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale
Visual analog scale | 3th week
  The Visual Analog Scale is a pain rating scale with the numbers 0. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale
Visual analog scale | 12th week
  The Visual Analog Scale is a pain rating scale with the numbers 0. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale
Range of Motion | 0( baseline)
  Shoulder ROM is measured using a universal protractor(goniometer). Shoulder ﬂection, extension, abduction, internal rotation and external rotation ranges are measured in the supine position.
Range of Motion | 3th week
  Shoulder ROM is measured using a universal protractor(goniometer). Shoulder ﬂection, extension, abduction, internal rotation and external rotation ranges are measured in the supine position.
Range of Motion | 12th week
  Shoulder ROM is measured using a universal protractor(goniometer). Shoulder ﬂection, extension, abduction, internal rotation and external rotation ranges are measured in the supine position.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 0( baseline)
  SPADI is a scale consisting of a total of 13 questions with 2 subscales: pain and disability. Total and all sub-parameter scores are evaluated on a 0-100 scale. A high score indicates increased pain and impaired shoulder function.
Shoulder Pain and Disability Index (SPADI) | 3th week
  SPADI is a scale consisting of a total of 13 questions with 2 subscales: pain and disability. Total and all sub-parameter scores are evaluated on a 0-100 scale. A high score indicates increased pain and impaired shoulder function.
Shoulder Pain and Disability Index (SPADI) | 12th week
  SPADI is a scale consisting of a total of 13 questions with 2 subscales: pain and disability. Total and all sub-parameter scores are evaluated on a 0-100 scale. A high score indicates increased pain and impaired shoulder function.
Modified Constant-Murley Score | 0( baseline)
  Modified Constant-Murley Score includes four parameters: pain, activities of daily living (ADL), active ROM and strength. The total score is evaluated on a 0-100 point scale by summing all sub-parameters. A low score reflects increased pain and impaired shoulder function for both sub-parameters and total score.
Modified Constant-Murley Score | 3th week
  Modified Constant-Murley Score includes four parameters: pain, activities of daily living (ADL), active ROM and strength. The total score is evaluated on a 0-100 point scale by summing all sub-parameters. A low score reflects increased pain and impaired shoulder function for both sub-parameters and total score.
Modified Constant-Murley Score | 12th week
  Modified Constant-Murley Score includes four parameters: pain, activities of daily living (ADL), active ROM and strength. The total score is evaluated on a 0-100 point scale by summing all sub-parameters. A low score reflects increased pain and impaired shoulder function for both sub-parameters and total score.
SF-36 | 0( baseline)
  Short-form health survey 36 (SF-36) contains 36 items that are used to evaluate the quality of life of patients with chronic pain. It measures eight different domains that address physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitation, and mental health. The score of each domain ranges from 0 (worse quality of life) to 100 (best quality of life). This assessment will be performed at pre-treatment, after 3 weeks of treatment and 12-week follow-up.
SF-36 | 3th week
  Short-form health survey 36 (SF-36) contains 36 items that are used to evaluate the quality of life of patients with chronic pain. It measures eight different domains that address physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitation, and mental health. The score of each domain ranges from 0 (worse quality of life) to 100 (best quality of life). This assessment will be performed at pre-treatment, after 3 weeks of treatment and 12-week follow-up.
SF-36 | 12th week
  Short-form health survey 36 (SF-36) contains 36 items that are used to evaluate the quality of life of patients with chronic pain. It measures eight different domains that address physical functioning, physical role limitation, pain, general health, vitality, social functioning, emotional role limitation, and mental health. The score of each domain ranges from 0 (worse quality of life) to 100 (best quality of life). This assessment will be performed at pre-treatment, after 3 weeks of treatment and 12-week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem KARACAY, assist prof, Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kirşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
participant data (IPD) will not available to other researchers.

REFERENCES:
- [Background] Sveistrup H, McComas J, Thornton M, Marshall S, Finestone H, McCormick A, Babulic K, Mayhew A. Experimental studies of virtual reality-delivered compared to conventional exercise programs for rehabilitation. Cyberpsychol Behav. 2003 Jun;6(3):245-9. doi: 10.1089/109493103322011524. PMID 12855079
- [Background] Lee SH, Yeh SC, Chan RC, Chen S, Yang G, Zheng LR. Motor Ingredients Derived from a Wearable Sensor-Based Virtual Reality System for Frozen Shoulder Rehabilitation. Biomed Res Int. 2016;2016:7075464. doi: 10.1155/2016/7075464. Epub 2016 Aug 23. PMID 27642600
- [Background] Gumaa M, Rehan Youssef A. Is Virtual Reality Effective in Orthopedic Rehabilitation? A Systematic Review and Meta-Analysis. Phys Ther. 2019 Oct 28;99(10):1304-1325. doi: 10.1093/ptj/pzz093. PMID 31343702